CLINICAL TRIAL: NCT01876602
Title: Feeling States and Heart Rates; A Translational Study
Brief Title: Test of an Intervention to Increase Physical Activity Among School Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Irvine (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Margaret Schneider, Principal Investigator, University of California, Irvine
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: DK088800; R01DK088800 (NIH)
Record Dates: First submitted 2013-06-10; First posted 2013-06-12 (Estimated); Last update posted 2018-05-15 (Actual); Status verified 2018-05

CONDITIONS: Obesity
Keywords: adolescents; exercise; fitness; school-based
MeSH Terms: conditions — Obesity; Motor Activity

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Exercise prescription (Experimental): Participants are given an exercise prescription in the form of a target heart rate range for exercising. The range is determined based on their personal preferences so that it is an intensity that feels "good".
  Interventions: Behavioral: feeling states exercise intervention
- traditional exercise (Active Comparator): participants are given an exercise prescription based on percent of vo2 peak
  Interventions: Behavioral: feeling states exercise intervention

INTERVENTIONS:
Behavioral: feeling states exercise intervention — exercise prescription based on intensity of exercise that feels good.

SUMMARY:
The specific aims of this study are to: 1) evaluate the impact of a novel intervention delivered via school-based physical education (PE) on adolescents who have a high sensitivity to exercise-induced negative affect; 2) determine whether adolescents' tendency to feel uncomfortable during exercise is a stable trait that persists even in the face of an intervention; and 3) compare and contrast three alternative methods of measuring adolescents' sensitivity to exercise-induced affect.

Healthy middle-school students who do not participate in team or individual competitive sports will be recruited and assessed to determine their existing predisposition toward exercise (i.e., "reluctant exercisers" and "latent exercisers"). The assessment will be conducted using three methods that have been used to measure individuals' propensity to experience positive affect in the face of a stimulus: 1) a pencil-and-paper assessment that measures tendency to respond to a challenge with positive affect; 2) electroencephalogram (EEG) to ascertain frontal cortical asymmetry; and 3) empirically assessed affective response to a standardized exercise task. Reluctant and latent exercisers will be assigned in equal numbers to one of two conditions. One condition will implement a PE-based intervention that differs from the traditional approach in that students will be instructed to exercise at an intensity that has been determined to elicit positive affect in that individual (based on baseline testing). In the other condition, students will be instructed to exercise at an intensity derived from standard formulas typically used in exercise prescriptions. It is hypothesized that the non-traditional approach will increase reluctant exercisers' enjoyment of PE and also their level of participation in physical activity outside of PE. The latter will be determined using portable monitors (accelerometers) worn at baseline, after the intervention, and again 1 year after the end of the intervention.

DETAILED DESCRIPTION:
This project addresses the current epidemic in obesity and physical inactivity among adolescents in the United States. The goal of the research is to develop effective ways of encouraging adolescents to become and remain physically active. In particular, this project is concerned with identifying adolescents who are reluctant to exercise because they have a high sensitivity to unpleasant feelings while exercising at higher intensities. Once identified, these adolescents can be targeted with an intervention that is designed to teach them to exercise at an intensity level that will generate pleasant feelings and therefore make it more likely that they will seek out opportunities to be physically active. The specific aims of this study are to: 1) evaluate the impact of a novel intervention delivered via school-based physical education (PE) on adolescents who have a high sensitivity to exercise-induced negative affect; 2) determine whether adolescents' tendency to feel uncomfortable during exercise is a stable trait that persists even in the face of an intervention; and 3) compare and contrast three alternative methods of measuring adolescents' sensitivity to exercise-induced affect.

Healthy middle-school students who do not participate in team or individual competitive sports will be recruited and assessed to determine their existing predisposition toward exercise (i.e., "reluctant exercisers" and "latent exercisers"). The assessment will be conducted using three methods that have been used to measure individuals' propensity to experience positive affect in the face of a stimulus: 1) a pencil-and-paper assessment that measures tendency to respond to a challenge with positive affect; 2) electroencephalogram (EEG) to ascertain frontal cortical asymmetry; and 3) empirically assessed affective response to a standardized exercise task. Reluctant and latent exercisers will be assigned in equal numbers to one of two conditions. One condition will implement a PE-based intervention that differs from the traditional approach in that students will be instructed to exercise at an intensity that has been determined to elicit positive affect in that individual (based on baseline testing). In the other condition, students will be instructed to exercise at an intensity derived from standard formulas typically used in exercise prescriptions. It is hypothesized that the non-traditional approach will increase reluctant exercisers' enjoyment of PE and also their level of participation in physical activity outside of PE. The latter will be determined using portable monitors (accelerometers) worn at baseline, after the intervention, and again 1 year after the end of the intervention.

This study is relevant to the prevention of type 2 diabetes in that it addresses the mechanisms of physical activity behavior change among adolescents. This developmental period is typically characterized by declining participation in physical activity, and thus represents a critical period for intervention. The results will increase understanding about why some adolescents remain active while others do not and will test a novel intervention that may be more effective among reluctant exercisers.

ELIGIBILITY:
Inclusion Criteria:

* Healthy
* not a member of a sports team
* right handed

Exclusion Criteria:

* no past head trauma
* not depressed

Ages: 10 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 140 (Actual)
Dates: Start 2011-04; Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Physical Activity | 1 year
  Participation in physical activity is assessing objectively (using activity monitors), by self-report, and indirectly via cardiorespiratory fitness.

SECONDARY OUTCOMES:
affective response to exercise | 1 year
  Affective response to exercise is assessed by measuring how participants feel during a standardized exercise task and by self-report of enjoyment of activity.

CONTACTS AND LOCATIONS:
Overall Officials: Margaret Schneider, PhD, Principal Investigator — University of California, Irvine
Locations (1):
- University of California at Irvine, Irvine, California, United States

REFERENCES:
- [Background] Schneider M, Schmalbach P, Godkin S. Impact of a personalized versus moderate-intensity exercise prescription: a randomized controlled trial. J Behav Med. 2017 Apr;40(2):239-248. doi: 10.1007/s10865-016-9776-0. Epub 2016 Aug 1. PMID 27481104
- [Derived] Schneider M. Intrinsic Motivation Mediates the Association Between Exercise-Associated Affect and Physical Activity Among Adolescents. Front Psychol. 2018 Jul 30;9:1151. doi: 10.3389/fpsyg.2018.01151. eCollection 2018. PMID 30104987
- [Derived] Schneider M, Schmalbach P. Affective Response to Exercise and Preferred Exercise Intensity Among Adolescents. J Phys Act Health. 2015 Apr;12(4):546-52. doi: 10.1123/jpah.2013-0442. Epub 2014 Apr 17. PMID 24770461